CLINICAL TRIAL: NCT00375791
Title: An Open-Label Phase II Study of the Safety and Efficacy of Perifosine Alone and in Combination With Dexamethasone for Patients With Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: Efficacy of Perifosine Alone and in Combination With Dexamethasone for Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 212
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2012-02

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — perifosine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perifosine daily (Experimental): Patients will take three 50 mg tablets of perifosine daily at bedtime with food. Patients will be examined every three weeks. If patients have no progression it is allowed to receive 8 cycles of perifosine
  Interventions: Drug: perifosine
- Perifosine daily + Dexa twice per week (Experimental): Patients will take three 50 mg tablets of perifosine daily at bedtime with food until progression. If progressive disease is confirmed by a second measurement at least one week later the patient will receive a combination of 20 mg twice per week dexamethasone (dexa) and 150 mg perifosine daily at bedtime.
  Interventions: Drug: perifosine; Drug: dexamethasone

INTERVENTIONS:
Drug: perifosine — 100 - 150 mg daily
  Other Names: D-21266; KRX-0401
Drug: dexamethasone — 20 mg twice weekly
  Other Names: decadron
  Arms: Perifosine daily + Dexa twice per week

SUMMARY:
This is a phase 2 study of perifosine in patients with multiple myeloma. Patients will receive perifosine 150 mg at bedtime (qhs) daily. Patients will be assessed by serum and/or urine-electrophoresis at least every 3 weeks.

DETAILED DESCRIPTION:
Treatment: Patients will take three 50 mg tablets of perifosine qhs daily with food. All patients should continue therapy unless disease progression is documented on two occasions at least 1 week apart. Progressing patients will have dexamethasone 20 mg twice per week added to the perifosine. Patients who experience toxicity may continue on treatment with doses delayed or reduced.

Evaluations: Serum and/or urine-electrophoresis will be evaluated for progression or response at 3 week intervals.

This study will enroll a total of up to 64 patients.

ELIGIBILITY:
Inclusion Criteria:

Major criteria:

1. Plasmacytomas on tissue biopsy.
2. Bone marrow plasmacytosis (> 30% plasma cells).
3. Monoclonal immunoglobulin spike on serum electrophoresis immunoglobulin G (IgG) > 3.5 g/dL or immunoglobulin A (IgA) > 2.0 g/dL; kappa or lambda light chain excretion > 1 g/day on 24 hour urine protein electrophoresis.

Minor criteria:

1. Bone marrow plasmacytosis (10 to 30% plasma cells)
2. Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
3. Lytic bone lesions
4. Normal immunoglobulin M (IgM) < 50 mg/dL, IgA < 100 mg/dL or IgG < 600 mg/dL.

Any of the following sets of criteria will confirm the diagnosis of multiple myeloma:

1. Any two of the major criteria.
2. Major criterion 1 plus minor criterion b, c or d.
3. Major criterion 3 plus minor criterion a or c.
4. Minor criteria a, b and c or a, b and d.

Exclusion Criteria:

1. Renal insufficiency (serum creatinine levels > 3 mg/dL).
2. Patients who present with either ALT or AST ≥ 2.5 X upper limit of normal.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
4. Concomitant therapy medications that include corticosteroids (except as indicated for other medical conditions, or up to 100 mgs of hydrocortisone as premedication for administration of certain medications or blood products) or other chemotherapy that is or may be active against myeloma, or therapy with chemotherapy within 3 weeks prior to Day 1. Nitrosoureas must be discontinued 6 weeks prior to Day 1.
5. Subjects with a hemoglobin < 8.0 g/dL.
6. Any condition, including laboratory abnormalities, that in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study.
7. Women of childbearing potential (WCBP) who are pregnant, or breast-feeding or men and women who are not using adequate contraception are excluded.
8. Plasma cell leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Response rate (the combined CR + PR + MR) with treatment perifosine | Every 3 weeks
  To determine the response rate (the combined Complete Response (CR) + Partial Response (PR) + Minor Response (MR) following treatment with perifosine in patients with multiple myeloma who have relapsed following Initial front-line therapy and are refractory to their most recent therapy.

SECONDARY OUTCOMES:
Response rate (CR + PR + MR) with combination therapy | Every 3 weeks
  To determine the response rate (CR + PR + MR) following treatment with combination therapy with perifosine plus dexamethasone in patients with multiple myeloma who have relapsed or were refractory to their most recent therapy before study enrollment, and failed to respond to or have relapsed following treatment with perifosine alone.
Assess the safety and tolerability of perifosine alone and in combination | Every 3 weeks
  To assess the safety and tolerability of perifosine alone and in combination with dexamethasone in patients with multiple myeloma.
Obtain correlative data in patients with multiple myeloma treated with perifosine and in combination | Every 3 weeks
  To obtain correlative data in patients with multiple myeloma treated with perifosine alone and in combination with dexamethasone.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Richardson, M.D, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - Investigative Site, Berkeley, California
  - Investigative Site, Duarte, California
  - Investigative Site, Atlanta, Georgia
  - Investigative Site, Chicago, Illinois
  - Investigative Site, Boston, Massachusetts
  - Investigative Site, Ann Arbor, Michigan
  - Investigative Site, Charlottesville, Virginia

REFERENCES:
- [Result] Blood (ASH Annual Meeting Abstracts) 2007 110: Abstract 1164 © 2007 American Society of Hematology